CLINICAL TRIAL: NCT02422784
Title: A Double-Blind, Randomized, Control Study to Examine the Effects of Vitamin D Fortification on Vitamin D Metabolite Profiles and Status in Vitamin D Insufficient Individuals.
Brief Title: Effects of Vitamin D Fortification on Vitamin D Metabolite Profiles and Status in Vitamin D Insufficient Individuals
Acronym: VITD-2013
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canada Manitoba Agri-Food Research and Development Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2013:045; B2013:045 (Other: University of Manitoba Biomedical Research Ethics Board)
Record Dates: First submitted 2015-02-11; First posted 2015-04-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-03

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D insufficient; rooibos tea; calcium
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Participants will be instructed to consume 240 mL of iced-tea daily for 6 weeks. The iced-tea beverages do not contain added sugar or artificial sweeteners. Beverages will be prepared fresh weekly and picked up by participants during their weekly study visits.
  Interventions: Dietary Supplement: Rooibos Iced-Tea (Control)
- Rooibos Tea - Vitamin D3 (Active Comparator): Participants will be instructed to consume 240 mL of iced-tea fortified with 1000 IU water-soluable vitamin D3 daily for 6 weeks. The iced-tea beverages do not contain added sugar or artificial sweeteners. Beverages will be prepared fresh weekly and picked up by participants during their weekly study visits.
  Interventions: Dietary Supplement: Rooibos Tea - Vitamin D3
- Rooibos Tea- Vitamin D3 & Calcium (Active Comparator): Participants will be instructed to consume 240 mL of Rooibos iced-tea fortified with 1000 IU of water-soluable vitamin D3 and 360 mg of calcium daily for 6 weeks. The iced-tea beverages do not contain added sugar or artificial sweeteners. Beverages will be prepared fresh weekly and picked up by participants during their weekly study visits.
  Interventions: Dietary Supplement: Rooibos Tea- Vitamin D3 & Calcium

INTERVENTIONS:
Dietary Supplement: Rooibos Iced-Tea (Control) — Participants will consume 240 mL of Rooibos iced-tea daily for 6 weeks. The iced-tea beverage will not contain any added sugar or artificial sweeteners. Beverages will be prepared fresh weekly and picked up by participants during their weekly study visits.
  Arms: Control
Dietary Supplement: Rooibos Tea - Vitamin D3 — Participants will consume 240 mL of Rooibos iced-tea fortified with 1000 IU of water soluable Vitamin D3 daily for 6 weeks. The iced-tea beverage will not contain any added sugar or artificial sweeteners. Beverages will be prepared fresh weekly and picked up by participants during their weekly study visits.
  Arms: Rooibos Tea - Vitamin D3
Dietary Supplement: Rooibos Tea- Vitamin D3 & Calcium — Participants will consume 240 mL of Rooibos iced-tea fortified with 1000 IU of water soluable Vitamin D3 and 360 mg of Calicum daily for 6 weeks. The iced-tea beverage will not contain any added sugar or artificial sweeteners. Beverages will be prepared fresh weekly and picked up by participants during their weekly study visits.
  Arms: Rooibos Tea- Vitamin D3 & Calcium

SUMMARY:
This is a cross-sectional study designed to compare plasma/serum and urine vitamin D metabolite profiles of vitamin D sufficient and insufficient individuals.

There are two phases of this study.

Phase 1 - Consented study participants will attend a screening visit and provide a fasting blood and urine sample. Those individuals who are vitamin D insufficient based on serum 25(OH)D concentrations will be invited to participate in Phase II

Phase II - is a double-blind, randomized, control study designed to examine vitamin D status in vitamin D insufficient individuals consuming a water-soluble form of vitamin D3. Eligible participants will be asked to consume one of three beverages: i) rooibos iced-tea (control); ii) rooibos iced-tea fortified with 1000 IU of water-soluble vitamin D3; or iii) rooibos iced-tea fortified with 1000 IU of water-soluble vitamin D3 and 360 mg calcium at 240 mL of iced-tea consumed daily for 6 weeks. Participants will attend 6 weekly visits following baseline and provide a fasting blood sample for assessment of serum 25(OH)D concentrations.

Objectives: 1) To investigate plasma/serum and urine vitamin D metabolite profiles in vitamin D sufficient and insufficient individuals; and 2) To determine the effects of vitamin D3 fortification on serum 25-dihydroxy-vitamin D [25(OH)D] concentrations, markers of vitamin D and calcium metabolism, and vitamin D metabolite profile in plasma/serum and urine of vitamin D insufficient individuals.

DETAILED DESCRIPTION:
Health individuals from the general public will be recruited into this cross-sectional study designed to compare plasma/serum and urine vitamin D metabolite profiles of those identified as vitamin D sufficient and insufficient individuals.

There are two objectives:

Objective 1: To investigate plasma/serum and urine vitamin D metabolite profiles in vitamin D sufficient and insufficient individuals; N=20 and will consist of 10 individuals identified as vitamin D insufficient and 10 individuals identified as vitamin D deficient individuals.

Objective 2: To determine the effects of vitamin D3 fortification on serum 25-dihydroxy-vitamin D [25(OH)D] concentrations, markers of vitamin D and calcium metabolism, and vitamin D metabolite profile in plasma/serum and urine of vitamin D insufficient individuals. N=45.

To achieve the objectives, the study will be conducted in two phases:

Phase 1 - Healthy males or females, ≥19 and ≤50 years of age, will be recruited from the general public. Consented study participants will provide a fasting blood and urine sample for the purpose of determination of vitamin D status (insufficient vs. deficient) based on serum 25(OH)D concentrations. Forty-five (45) individuals identified as vitamin D insufficient (having a serum 25(OH)D concentration ≥30 and ≤75 nmol/L) will proceed to phase II. A N=20 (10 vitamin D insufficient and 10 vitamin D deficient) will also be identified to satisfy objective 1.

Phase II - is a double-blind, randomized, control study designed to examine vitamin D status in vitamin D insufficient individuals consuming a water-soluble form of vitamin D3. Eligible participants will randomized to consume one of three beverages: i) rooibos iced-tea (control); ii) rooibos iced-tea fortified with 1000 IU of water-soluble vitamin D3; or iii) rooibos iced-tea fortified with 1000 IU of water-soluble vitamin D3 and 360 mg calcium at 240 mL of iced-tea consumed daily for 6 weeks. Both researchers and participants will be blinded to the beverage group assigned to each participant. Participants will then attend 6 weekly visits following the baseline visit to provide fasting blood samples for assessment of serum 25(OH)D concentrations.

Analysis of intact-PTH, alkaline-phosphatase, calcium, phosphorus, CRP, TAP and vitamin D metabolite profile and a urine sample will also be obtained for assessment of N-telopeptide and vitamin D metabolite profile will also occur at Baseline and Week 6. Fasting blood samples collected at week 3 will be used for additional assessment of serum alkaline phosphatase, calcium and phosphorus. A 3-day Food Record will be provided at week 3.

Vitamin D insufficient participants will be stratified according to their serum 25(OH)D concentrations (≥30 and ≤50, or >50 and ≤75 nmol/L) after screening and prior to the beverage study to ensure that a range of lower and higher serum 25(OH)D concentrations are represented in each beverage group.

ELIGIBILITY:
Inclusion Criteria:

A. Inclusion Criteria for Objective 1 (Part One):

1. Adult volunteers, male or female, between 19 and 50 years of age;
2. Body mass index (BMI) ≥20 and ≤30 kg/m2 (normal to overweight);
3. Must be on a stable regime for the past three months, if taking vitamin and mineral/dietary/herbal supplements; and
4. Willing to provide informed consent.

B. Inclusion Criteria for Objective 2 (Part Two):

1. Adult volunteers, male or female, between 19 and 50 years of age;
2. Body mass index (BMI) ≥20 and ≤30 kg/m2 (normal to overweight);
3. Must be on a stable regime for the past three months, if taking vitamin and mineral/dietary/herbal supplements;
4. Vitamin D insufficient (serum 25(OH)D concentrations ≥30 and ≤75 nmol/L);
5. Willing to comply with protocol requirements; and
6. Willing to provide informed consent.

Exclusion Criteria:

1. Take a vitamin D or calcium supplement within the last three months before the start date of the study, or during the study;
2. History of vitamin D deficiency (serum 25(OH)D concentration <30 nmol/L);
3. History of hypocalcaemia;
4. Presence of a clinically diagnosed disease affecting the circulatory, respiratory, immune, skeletal, urinary, muscular, endocrine, digestive, nervous or reproductive system that requires medical treatment;
5. Taking any medication (with the exception of birth control);
6. Daily consumption of more than three servings of dairy products;
7. Undergone significant sun exposure one month before start date of the study;
8. Use or have used a tanning booth one month before start date of the study, or during the study;
9. Plan to travel to a sunny climate during the study;
10. Currently smoking or have smoked within the last six months before start date of the study, or during the study;
11. Have allergies to tea products;
12. Pregnant or lactating; and
13. Consume excessive alcohol (>10 drinks/week for women, >15 drinks/week for men).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Plasma/Serum and Urine Vitamin D Metabolite Profiles of Vitamin D Sufficient and Insufficient Individuals | Screening Visit (Day 0) - Phase 1
  To investigate plasma/serum and urine vitamin D metabolite profiles in vitamin D sufficient and insufficient individuals.
The Effects of Vitamin D Fortification on Serum 25(OH)D in Vitamin D Insufficient Individuals. | 6 Weeks (Phase II)
  To determine the effects of 6 weeks of vitamin D3 fortification on serum 25-dihydroxy-vitamin D [25(OH)D] concentrations of vitamin D insufficient individuals.

SECONDARY OUTCOMES:
The Effects of Vitamin D3 Fortification on markers of vitamin D of vitamin D insufficient individuals | 6 Weeks (Phase II)
  To determine the effects of 6 weeks of vitamin D3 fortification on markers of vitamin D in plasma/serum and urine of vitamin D insufficient individuals.
The Effects of vitamin D3 Fortification on calcium metabolism of Vitamin D Insufficient Individuals. | 6 Weeks (Phase II)
  To determine the effects of 6 weeks of vitamin D3 fortification on calcium metabolism in plasma/serum and urine of vitamin D insufficient individuals.
The Effects of Vitamin D3 Fortification on Vitamin D Metabolite Profile of Vitamin D Insufficient Individuals. | 6 Weeks (Phase II)
  Determine the effects of vitamin D3 fortification on the vitamin D metabolite profile in plasma/serum and urine of vitamin D insufficient individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital, Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Calvo MS, Whiting SJ, Barton CN. Vitamin D fortification in the United States and Canada: current status and data needs. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1710S-6S. doi: 10.1093/ajcn/80.6.1710S. PMID 15585792
- [Background] Tangpricha V, Koutkia P, Rieke SM, Chen TC, Perez AA, Holick MF. Fortification of orange juice with vitamin D: a novel approach for enhancing vitamin D nutritional health. Am J Clin Nutr. 2003 Jun;77(6):1478-83. doi: 10.1093/ajcn/77.6.1478. PMID 12791627
- [Background] Ding S, Schoenmakers I, Jones K, Koulman A, Prentice A, Volmer DA. Quantitative determination of vitamin D metabolites in plasma using UHPLC-MS/MS. Anal Bioanal Chem. 2010 Sep;398(2):779-89. doi: 10.1007/s00216-010-3993-0. Epub 2010 Jul 14. PMID 20628873
- [Background] Luque de Castro MD, Fernandez-Romero JM, Ortiz-Boyer F, Quesada JM. Determination of vitamin D3 metabolites: state-of-the-art and trends. J Pharm Biomed Anal. 1999 Jun;20(1-2):1-17. doi: 10.1016/s0731-7085(99)00027-8. PMID 10704005
- [Background] Stalmach A, Mullen W, Pecorari M, Serafini M, Crozier A. Bioavailability of C-linked dihydrochalcone and flavanone glucosides in humans following ingestion of unfermented and fermented rooibos teas. J Agric Food Chem. 2009 Aug 12;57(15):7104-11. doi: 10.1021/jf9011642. PMID 19534535
- See also: Canadian Centre for Agri-Food Research in Health and Medicine — http://www.ccarm.ca